CLINICAL TRIAL: NCT02407652
Title: Cognitive Control Training as a Preventive Intervention for Depression: A Double-blind Randomized Controlled Trial Study
Brief Title: Cognitive Control Training for Remitted Depressed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B/13808/01-CCT-003
Record Dates: First submitted 2015-03-10; First posted 2015-04-03 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Major Depression in Remission

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cognitive control training (Experimental): internet-delivered, 2 weeks
  Interventions: Behavioral: Cognitive Control Training
- low cognitive load training (Active Comparator): internet-delivered, 2 weeks
  Interventions: Behavioral: Low Cognitive Load Training

INTERVENTIONS:
Behavioral: Cognitive Control Training — 10 adaptive Paced Auditory Serial Addition Task (PASAT) sessions, 400 trials each
  Arms: cognitive control training
Behavioral: Low Cognitive Load Training — 10 low cognitive load sessions, 400 trials each
  Arms: low cognitive load training

SUMMARY:
The purpose of this study is to explore the effectiveness of an internet-delivered cognitive control training as a preventive intervention for remitted depressed patients.

DETAILED DESCRIPTION:
Prospective studies have linked impaired cognitive control to increased cognitive vulnerability for future depression. Importantly, experimental studies indicate that cognitive control training can be used to reduce rumination and depressive symptomatology in MDD samples. Furthermore, studies exploring the potential of cognitive control training in at-risk undergraduate students indicate that cognitive control training has beneficial effects on rumination, an important vulnerability factor for depression. Provided that remitted depressed patients form a high-risk group for developing future depressive episodes, the current study will explore whether internet-delivered cognitive control training can be used to reduce vulnerability for future depression in remitted depressed patients. The investigators will explore effects on depressive symptomatology, (mal-)adaptive emotion regulation (directly following training and at 3 months follow-up), and indices of functioning (at 3 months follow-up).

ELIGIBILITY:
Inclusion Criteria:

* History of ≥ 1 depressive episode(s)
* Currently in stable full or partial remission (≥ 6 months)

Exclusion Criteria:

* Major depressive disorder (MDD; current)
* Bipolar disorder (current and/or previous)
* Psychotic disorder (current and/or previous)
* Neurological impairments (current and/or previous)
* Excessive substance abuse (current and/or previous)
* No other comorbid disorders (current)
* No ongoing psychotherapeutic treatment (maintenance treatment is allowed, but with a frequency less than once / 3 weeks)
* Use of antidepressant medication is allowed if kept at a constant level

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in depressive rumination from baseline to the post-training assessment and follow-up (RRS) | baseline, 2 weeks, 3 months
  Assessed using the Ruminative Response Scale (RRS)
Change in depressive symptomatology from baseline to the post-training assessment and follow-up (BDI-II) | baseline, 2 weeks, 3 months
  Assessed using the Beck Depression Inventory (BDI-II)

SECONDARY OUTCOMES:
(mal-)Adaptive cognitive emotion regulation (CERQ) | baseline, 2 weeks, 3 months
  Assessed using the Cognitive Emotion Regulation Questionnaire (CERQ)
Quality of Life (QLDS) | baseline, 3 months
  Assessed using the Quality of Life in Depression Scale (QLDS)
Disability (WHODAS 2.0) | baseline, 3 months
  Assessed using the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0)
Resilience (RS) | baseline, 3 months
  Assessed using the Resilience Scale (RS)
Remission from depression (RDQ) | baseline, 3 months
  Assessed using the Remission of Depression Questionnaire (RDQ)

OTHER OUTCOMES:
Behavioral measure for cognitive control ((non-adaptive) PASAT) | baseline, 2 weeks, 3 months
  Assessed using the (non-adaptive) PASAT
Self-reported cognitive control (BRIEF-A) | baseline, 2 weeks, 3 months
  Assessed using the Behaviour Rating Inventory of Executive Function Adult Version (BRIEF-A)

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Koster, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

REFERENCES:
- [Derived] Hoorelbeke K, Koster EHW. Internet-delivered cognitive control training as a preventive intervention for remitted depressed patients: Evidence from a double-blind randomized controlled trial study. J Consult Clin Psychol. 2017 Feb;85(2):135-146. doi: 10.1037/ccp0000128. Epub 2016 Jun 30. PMID 27362792
- [Derived] Hoorelbeke K, Faelens L, Behiels J, Koster EH. Internet-delivered cognitive control training as a preventive intervention for remitted depressed patients: Protocol for a randomized controlled trial. BMC Psychiatry. 2015 Jun 9;15:125. doi: 10.1186/s12888-015-0511-0. PMID 26055122